CLINICAL TRIAL: NCT06863714
Title: Effect Of Peritonsillar Bupivacaine Infiltration on The Development of Postoperative Emergence Delirium After Tonsillectomy In Children: A Randomized, Double-Blind, Controlled Study
Brief Title: Peritonsillar Bupivacaine Infiltration After Tonsillectomy In Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hacer Sebnem Turk, associate professor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: turk-24
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Post Operative Delirium; Post Operative Pain
Keywords: Emergence Delirium; Tonsillectomy; Bupivacaine; Infiltration Analgesia; Postoperative Pain
MeSH Terms: conditions — Emergence Delirium; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Peritonsillar injection was superficially administered to the superior and inferior peritonsillar regions in a volume of 2-5 ml. A 23 Gouge needle syringe was used for injection. A 0.5% Bupivacaine was administered at a dose of 1 mg/kg (maximum dose of 25 mg)
  Interventions: Drug: peritonsillar bupivacaine injection
- group B (No Intervention): no intervetion

INTERVENTIONS:
Drug: peritonsillar bupivacaine injection — Peritonsillar injection was superficially administered to the superior and inferior peritonsillar regions in a volume of 2-5 ml. A 23 Gouge needle syringe was used for injection. A 0.5% Bupivacaine was administered at a dose of 1 mg/kg (maximum dose of 25 mg)
  Arms: Group A

SUMMARY:
To evaluate the effect of peritonsillar bupivacaine infiltration on the development of postoperative delirium in pediatric patients undergoing tonsillectomy or adenotonsillectomy.

DETAILED DESCRIPTION:
Postoperative emergence delirium (ED) is an important clinical condition characterized by crying, irritability and severe restlessness in subjects recovering from anesthesia. ED is more common in children than in adults. Among the types of surgery, the ED is common in ENT surgery in which the prevalence was reported between 13%-26%. The adenotonsillectomy, which is a common ENT procedure carry a high risk for development of ED.

The ED can cause the child recovering from anesthesia to harm himself/herself and the surgical site and may cause parents to question the quality of anesthesia. It is associated with postoperative increased morbidity. Several anesthetic strategies exists (intranasal premedication, deep versus awake removal of the laryngeal mask, different intravenous anesthetic combinations) in the literature in order to prevent delirium. Local anesthetic application as xylocaine was shown to reduce the postoperative pain and ED. In addition it is generally accepted that that postoperative ED can be reduced with good analgesia.

Local infiltration of peritonsillar fossa with various local anesthetics, steroids etc. is an established technique for relieving the postoperative pain. Bupivacaine as a long-acting local anesthetic is widely used for local infiltration anesthesia. It is a safe technique and several comparative studies exists in the literature on efficacy. A few number of studies exists that evaluates the relationship between effective pain control and postoperative ED development in children with regional anesthesia applications. However, in English literature we could not find a study on the effect of local infiltration of peritonsillar fossa on development of ED in subjects who underwent tonsillectomy/adenotonsillectomy operations.

The aim of this study is to evaluate the effect of peritonsillar bupivacaine infiltration on the development of postoperative delirium in pediatric patients undergoing tonsillectomy/adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient have adenotonsillectomy
* age 3-7 years
* ASA-1

Exclusion Criteria:

* active infection,
* bleeding-coagulation disorder,
* neuropsychiatric disorder,
* bupivacaine hypersensitivity,
* postoperative delirium history,
* history of surgery for different reasons within 1 year,
* history of long-term hospitalization,
* chronic disease,
* chronic pain condition
* chronic analgesic use

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Pediatric Emergence Delirium Scale | PAED scores were measured at the beginning, 5th, 10th, 20th, 30th and 60th minutes in the postoperative recovery unit.
  This scale system was created to evaluate the severity of delirium in children patients. In thİs scale system, patients are graduated between 0 and 20 points. A score of 0 reveals there are no delirium findings, and a score of 20 reveals there is a severe delirium.

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability | FLACC scores were measured at the beginning, 5th, 10th, 20th, 30th and 60th minutes in the postoperative recovery unit.
  The Face, Legs, Activity, Cry and Consolability score is a scoring system created to evaluate the severity of pain in children in the postoperative period. The lowest score of 0 represents no pain, while a score of 10 indicates high pain severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No